CLINICAL TRIAL: NCT01768026
Title: A Prospective, Longitudinal Assessment of Disease Severity in Subjects With Dystrophic Epidermolysis Bullosa (DEB)
Brief Title: Prospective, Longitudinal Natural History Study in Dystrophic Epidermolysis Bullosa
Status: Withdrawn | Type: Observational
Sponsor: Lotus Tissue Repair, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DEB-101-12
Record Dates: First submitted 2013-01-10; First posted 2013-01-15 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-02

CONDITIONS: Dystrophic Epidermolysis Bullosa
Keywords: Dystrophic Epidermolysis Bullosa; Type VII Collagen; QOL Evaluation in Epidermolysis Bullosa; Instrument for Scoring Clinical Outcomes for Research of Epidermolysis Bullosa; Birmingham Epidermolysis Bullosa Severity Score
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Subjects diagnosed with Dystrophic Epidermolysis Bullosa

SUMMARY:
The objective of this study is to characterize the extent and severity of disease in subjects with DEB and the progression of disease over a timeframe relevant to interventional studies. The data from this study will be used to inform the study design and address statistical considerations of future treatment protocols.

DETAILED DESCRIPTION:
This is a prospective, multicenter, multinational, longitudinal assessment of disease severity in subjects with DEB. Subjects with either dominant or recessive DEB (dominant dystrophic epidermolysis bullosa (DDEB) and recessive dystrophic epidermolysis bullosa (RDEB), respectively) will be assessed four times over a one year period: upon enrollment, and at 1 to 2 weeks and 6 and 12 months after enrollment. All subjects with either DDEB or RDEB that meet the study entry criteria will be offered participation in the study, provided they can be accommodated within the anticipated study timeline. In addition to their usual clinic assessment, subjects will have a quantitative evaluation of skin involvement and will be asked to fill out questionnaires that measure among other things disease severity, QOL, pain, pruritus, and medical and family histories.

ELIGIBILITY:
Eligibility Criteria

* Subjects of any age (newborns included) may participate
* Subjects over 18 years of age and parent(s)/legal guardian(s) of subjects <18 years of age must provide written informed consent prior to participating in the study and informed assent will be obtained from minors at least 7 years of age
* Subjects must have a documented diagnosis of DEB based on clinical presentation and either skin biopsy results showing an absence or reduction in C7 or anchoring fibrils or genetic analysis showing a mutation in collagen, type VII, alpha 1 (Col7A1); alternatively, subjects must have a clinical diagnosis of DEB and a documented diagnosis of DEB (as above) in a first degree relative
* No experimental systemic therapy for DEB including, but not limited to, bone marrow transplantation, systemic immune suppression, or experimental therapies that involve live cells which have the potential for systemic spread such as gene transfer, stem cell infusions or other cell type injections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected from clinical sites with interdisciplinary clinics for Dystrophic Epidermolysis Bullosa
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Characterize the progression of disease severity in subjects with DEB over 6 - 12 months. | One year period
  Disease severity and its impact on quality of life and function will be investigated over a one year period at the following timepoints: upon enrollment, and at 1 to 2 weeks and 6 and 12 months after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Hal Landy, MD, Study Director — Lotus Tissue Repair, Inc.
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

REFERENCES:
- See also: Dystrophic Epidermolysis Bullosa Research Association of America (DEBRA) — http://www.debra.org/
- See also: EB Care Patient Reported Registry — https://ebcare.patientcrossroads.org/
- See also: Lotus Tissue Repair, Inc. — http://www.lotustissuerepair.com/
- See also: Dystrophic Epidermolysis Bullosa Research Association International — http://www.debra-international.org/homepage.html